CLINICAL TRIAL: NCT05246956
Title: Investigation of the Effect of Intradialytic Exercise on Functional Capacity and Quality of Life in Hemodialysis Patients
Brief Title: Investigation of the Effect of Intradialytic Exercise on Functional Capacity,Quality of Life in Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Medipol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Intradialytic Exercise
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2021-06

CONDITIONS: Renal Disease
Keywords: intradialytic exercise; chronic kidney disease; quality of life; depression; functional capacity
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic; Depression

STUDY DESIGN:
Intervention Model Description: experimental group control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intradialytic exercise in hemodialysis patients ( Experimental Group) (Experimental): Intradialytic exercise group
  Interventions: Other: Intradialytic exercise
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Other: Intradialytic exercise — Intradialytic exercise group
  Arms: Intradialytic exercise in hemodialysis patients ( Experimental Group)

SUMMARY:
Chronic renal failure (CKD) is defined as a chronic, progressive degeneration in the kidney's fluid-electrolyte balance and metabolic-endocrine functions as a result of the glomerular filtration rate (GFR) falling below 60 ml/min/1.73 m², regardless of the etiology of the kidney disease. CRF is divided into five stages according to the glomerular filtration rate. Stage V is end-stage renal disease (ESRD), a life-threatening condition in which GFR falls below 15 ml/min/1.73 m2. ESRD patients have to receive dialysis [hemodialysis (HD), peritoneal dialysis (PD)] or kidney transplantation (Tx) under the name of renal replacement therapies (RRT) in order to survive and to support the metabolic hemostatic function of the kidney. Although the majority of ESRD patients survive on dialysis, their quality of life and functional capacity are reduced due to uremic cardiomyopathy, cardiovascular diseases, anemia, diabetes mellitus, bone diseases, deconditioning, fatigue, weakness, inactivity and accompanying psychological problems. In addition, due to the burden of chronic disease and the necessity of being dependent on machinery, patients are also faced with the risk of losing their job, addiction in daily life activities, depression, anxiety, changes in body image, financial problems, sexual problems, social isolation, mortality and hospitalization.

Intradialytic exercise (IDE) is defined as exercise training performed during the hemodialysis session to increase the patient's strength and endurance and thus target various physiological and psychosocial parameters. Patients' choice of exercise depends on individual factors such as medical history, physical capacity, and transportation options, which are associated with cost and overall preferences. In this context, exercise programs during dialysis and at home are more preferred by patients due to the lack of transfer problems and loss of time. The exercise rehabilitation program to be chosen should also have features such as being practical, low cost and sustainable for patients receiving dialysis. Intradialytic exercise is a common recommendation to encourage patients to be physically active. Previous studies have shown that intradialytic exercise can reduce the severity of fatigue, improve sleep quality, increase exercise tolerance, improve life He claimed that it was effective in improving the quality of life and even improving the psychological state. Patients typically undergo two or three hemodialysis sessions per week, with each session lasting approximately 4 hours. As many patients maintain bed rest during hemodialysis sessions, intradialytic exercise can be a potentially useful approach to improve their health without spending extra time in the interdialytic period. Although exercise variety is limited during hemodialysis sessions, intradialytic exercise maximizes the use of HD time. In addition, intradialytic exercise has been reported to increase patient compliance. However, conflicting data on the effects of intradialytic exercise have been reported. Intradialytic exercise (IDE) is not yet a routine practice for hemodialysis patients, an important reason is the lack of guidelines to support it. Intradialytic exercise is rarely given as standard of care, although numerous small studies have demonstrated the multiple benefits and safe practice of intradialytic exercise training for patients with end-stage renal disease.

The aim of our study is to investigate the effect of intradialytic exercises on functional capacity and quality of life, although it is known that it can be done without spending extra time and is more preferred by patients, which is not routinely applied and needs more studies on its effects.

ELIGIBILITY:
Inclusion Criteria:

* Having stage 5 (ESRD) CRF according to GFR
* Being between 20-80 years old
* Ability to read and write
* Being cooperative
* Dialysis treatment for at least three months
* Willingness to participate in the research

Exclusion Criteria:

* History of myocardial ischemia in the last 6 months
* Uncontrolled diabetes mellitus and hypertension
* heart failure
* Having a malignant disease,
* Having mental retardation,
* illiteracy,
* Not being cooperative
* Having neurological or orthopedic disability.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
6 min walking test | 6 minute
Kidney Disease Quality of Life-36 Scale | 10 minute

SECONDARY OUTCOMES:
Beck Depression Inventory | 5 minute
Visual Analog Scale | 1 minute
  Fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Özal Keleş, Principal Investigator — Student
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No